CLINICAL TRIAL: NCT02035020
Title: A Phase IIa Clinical Trial to Test the Safety and Efficacy of Interferon Gamma Treatment in Elevating Frataxin Levels in Friedreich's Ataxia (FRDA) Patients
Brief Title: A Phase IIa Trial to Test Safety and Efficacy Interferon Gamma Treatment in Elevating Frataxin Levels in FRDA Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Carlo Casali, Professor, Azienda Policlinico Umberto I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIFT/1
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Friedreich Ataxia
Keywords: frataxin, gamma interferon, Friedreich ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gamma interferon (Experimental): IFN gamma 1b (Immukin ®) will be administered by subcutaneous route at day 0, 14 and 28 at a dose of 100, 150 and 200 ug respectively.
  Interventions: Drug: gamma interferon

INTERVENTIONS:
Drug: gamma interferon — IFN gamma 1b (Immukin ®) will be administered by subcutaneous route at day 0, 14 and 28 at a dose of 100, 150 and 200 ug respectively.
  Other Names: Imukin

SUMMARY:
The primary objective of this study is to investigate whether the treatment with IFN gamma can induce significant accumulation of frataxin in FRDA patients, a possibility suggested by pre-clinical evidence in an animal model of the disease.

DETAILED DESCRIPTION:
This is a Phase 2 clinical trial. A total of 10 FRDA patients will be recruited All subjects will be treated with a dose of 100-150-200-micrograms of IFN gamma 1b (Imukin®) subcutaneously, with an interval of 14 days, for a total of 3 injections.

ELIGIBILITY:
Inclusion Criteria:

1. FRDA patients should have their diagnosis genetically confirmed.
2. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
3. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
4. Male and/or female subjects between the ages of > 18 and < 45 years

   -

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Significant concurrent medical conditions at the time of screening or baseline visit, including, but not limited to, the following:

   * Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, GI, endocrine, pulmonary, immunologic, or local active infection/infectious illness) that, in the investigator's judgment, will substantially increase the risk to the subject if he or she participates in the study.
   * Class III or IV congestive heart failure as defined by the New York Heart Association.
   * Acute coronary syndrome (eg, myocardial infarction, unstable angina pectoris) and any history of significant cerebrovascular disease within 24 weeks before screening.
3. Presence of a transplanted organ.
4. Previous assumption of IFN gamma 1b.
5. Abnormality in any of the below hematology or chemistry profile values at screening:

   * Positive hepatitis B surface antigen (HBsAg), Total hepatitis B core antibody (HBcAb; also called anti HBc), and/or hepatitis C antibody (HCVAb) with confirmation by hepatitis C virus ribonucleic acid (HCV RNA).
   * ALT/AST levels > or = 1.5X ULN.
   * Total bilirubin level > or = 1.5 times the ULN.
   * Hemoglobin level < or = 80 gL (8.0 g/dL).
   * Platelet count < or = 100 x 109/L (100,000 cells/mm³) or > or = 1000 x 109/L (1,000,000 cells/mm³).
   * White blood cell count < or = 3.5 x 109/L (3500 cells/mm³).
   * Absolute neutrophil count (ANC) <2000 cells/mm³.
   * Serum creatinine level > or = 177 μmol/ L (2 mg/dL).
   * Glycosylated hemoglobin (HbA1c >10%).
6. Current or history of serious psychiatric disorder or alcohol or drug abuse.
7. Participation in other studies within 30 days before screening and/or during study participation.
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or ability to comply with study procedures, investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

   -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07-30 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Change in cellular frataxin | 24 hours and 7 days from each study drug administration
  The primary endpoint is to test the increase of cellular frataxin after treatment with IFN gamma. Quantitation of cellular frataxin will be performed after 24 hours and 7 days from each study drug administration

SECONDARY OUTCOMES:
Safety Blood sample | day 0-14-28-35
  Secondary endpoint is the safety and tolerability of IFN gamma in FRDA patients. The on treatment adverse events and withdrawals due to adverse effects will be reported. Any subject who receives at least 1 dose of investigational product will be included in the evaluation for safety

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Casali, MD, Principal Investigator — Policlinico Umberto I°
Locations (1):
- Policlinico Umberto I°, Rome, Italy/Rome, Italy

REFERENCES:
- [Background] Tomassini B, Arcuri G, Fortuni S, Sandi C, Ezzatizadeh V, Casali C, Condo I, Malisan F, Al-Mahdawi S, Pook M, Testi R. Interferon gamma upregulates frataxin and corrects the functional deficits in a Friedreich ataxia model. Hum Mol Genet. 2012 Jul 1;21(13):2855-61. doi: 10.1093/hmg/dds110. Epub 2012 Mar 23. PMID 22447512